CLINICAL TRIAL: NCT03954730
Title: Comparison Of Eccentric Training And Active Release Technique On Quadriceps Muscle In Patients With Dynamic Hip Screw
Brief Title: Eccentric Training Versus Active Release Technique On Quadriceps In Patients With Dynamic Hip Screw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Qurat-ul-ain Saeed
Record Dates: First submitted 2019-05-16; First posted 2019-05-17 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Hip Surgery
Keywords: Eccentric training; Active Release Technique

STUDY DESIGN:
Intervention Model Description: There will be two treatment groups of participants, One group will be trained on eccentric graded protocol whereas the other will receive active release technique of quadriceps.
Who Masked: Participant
Masking Description: Sealed envelope method is used to randomly assign participants into two groups. The therapist will know about the treatment but patient is not aware of treatment type.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric Training Group (Experimental): Eccentric training will be performed for quadriceps muscle along with strengthening protocol taken from Clinical Guidelines of NHS for post operative Dynamic Hip Screw rehabilitation.
  Interventions: Other: Eccentric Training
- Active Release Technique Group (Active Comparator): Active release technique will be performed for quadriceps muscle along with strengthening protocol taken from Clinical Guidelines of NHS for post operative Dynamic Hip Screw rehabilitation.
  Interventions: Other: Active Release Technique

INTERVENTIONS:
Other: Eccentric Training — First session will be performed 24 hours after pre-training tests i.e. on 4th post- operative day and subsequent sessions will be performed with lapse of 48 hours. During pre-testing, weight for the eccentric training will be determined using Standardized Brzycki formulas for lower limb. Participants will perform one set of 10 repetitions with selected weight. Intensity will be increased every week by decreasing the time of performance. Volume will be increased by increasing one set after two weeks. Eccentric training will be performed in sitting position on dynamic constant external resistance equipment.After session, patient will perform strengthening of quadriceps muscle as per clinical practice guidelines of National Health Service (UK).
  Arms: Eccentric Training Group
Other: Active Release Technique — Isometric Quadriceps' contractions against therapist's resistance lasting for 10 seconds will be performed by the patient in inner range of knee extension and after relaxing; actively perform maximum full knee flexion. Patient will perform extension at knee joint again; when reaches the innermost range, therapist will apply pressure on deep fascia either through knuckles/fingers or forearm in the direction towards the hip joint and patient is asked to perform knee flexion simultaneously. The procedure is applied onto vastus lateralis, rectus femoris and vastus intermedialis thrice in a session. After session, patient will perform strengthening of quadriceps muscle as per clinical practice guidelines of National Health Service (UK).
  Arms: Active Release Technique Group

SUMMARY:
This study will compare the effects of Eccentric training and Strength training with priory applied Active Release Technique on Quadriceps muscle in post operative patients of Dynamic Hip screw. Participants would be equally divided into two groups each receiving specific type of protocol besides standard post operative protocol of Dynamic Hip screw

DETAILED DESCRIPTION:
The study is Randomized Control Trial, being conducted at Fauji Foundation Hospital Rawalpindi .This study will compare the effects of two techniques addressing the contractile as well as non-contractile element of Quadriceps in early phase of Rehabilitation.

Sample size of 18 was calculated using software Epitool with 95% confidence interval and 80% power. Individuals of selected population will be randomly allocated as 9 in Eccentric group and 9 in Active Release Technique group by sealed enveloped method.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-65 years
* Patient with stable vitals on 3rd post-operative day
* Postero-Lateral Hip surgical approach

Exclusion Criteria:

* History of prior fracture
* History of fall
* Multiple fractures
* Cognitive impairment (Score ˂26 on Montreal cognitive assessment)
* Co-morbid disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline
  Numeric Pain Rating Scale (NPRS) is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Numeric Pain Rating Scale (NPRS) | post 6th week
  Numeric Pain Rating Scale (NPRS) is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Knee Range of Motion (ROM) | Baseline
  To assess Knee range of motion (ROM), Goniometer will be use to measure knee range of motion in flexion & extension. Participants will be seated upright and asked to actively move their knee in each direction.
Knee Range of Motion (ROM) | post 6th week
  To assess Knee range of motion (ROM), Goniometer will be use to measure knee range of motion in flexion & extension. Participants will be seated upright and asked to actively move their knee in each direction.

SECONDARY OUTCOMES:
Modified Harris Hip score(MHHS) | Baseline
  The modified Harris hip score (MHHS) is used to assess functional outcomes of hip joint. It is scored from 0 (worst functional outcome and maximum pain) to 100 points (best functional outcome and least pain).
Modified Harris Hip score(MHHS) | post 6th week
  The modified Harris hip score (MHHS) is used to assess functional outcomes of hip joint. It is scored from 0 (worst functional outcome and maximum pain) to 100 points (best functional outcome and least pain).

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amjad M, Akram R, Zaman AU, Ahmad I, Aziz A. Frequency and Causes of Failure of Dynamic Hip Screw Fixation for Interochanteric Fracture. PAKISTAN JOURNAL OF MEDICAL & HEALTH SCIENCES. 2016;10(3):734-40.
- [Background] Mue D, Salihu M, Awonusi F. Clinical Outcome Following Treatment Of Pertrochanteric Fractures With Dynamic Hip Screw In A Nigerian Rehabilitation Hospital. Journal of Dental and Medical Sciences. 2014;13(10):56-62.
- [Background] Carneiro MB, Alves DP, Mercadante MT. Physical therapy in the postoperative of proximal femur fracture in elderly. Literature review. Acta Ortop Bras. 2013 May;21(3):175-8. doi: 10.1590/S1413-78522013000300010. PMID 24453665
- [Background] Briggs RA, Houck JR, LaStayo PC, Fritz JM, Drummond MJ, Marcus RL. High-Intensity Multimodal Resistance Training Improves Muscle Function, Symmetry during a Sit-to-Stand Task, and Physical Function Following Hip Fracture. J Nutr Health Aging. 2018;22(3):431-438. doi: 10.1007/s12603-017-0977-1. PMID 29484358
- [Background] Briggs RA, Houck JR, Drummond MJ, Fritz JM, LaStayo PC, Marcus RL. Muscle Quality Improves with Extended High-Intensity Resistance Training after Hip Fracture. J Frailty Aging. 2018;7(1):51-56. doi: 10.14283/jfa.2017.31. PMID 29412443
- [Background] Hedayatpour N, Izanloo Z, Falla D. The effect of eccentric exercise and delayed onset muscle soreness on the homologous muscle of the contralateral limb. J Electromyogr Kinesiol. 2018 Aug;41:154-159. doi: 10.1016/j.jelekin.2018.06.003. Epub 2018 Jun 6. PMID 29902705